CLINICAL TRIAL: NCT05668832
Title: Bioavailability of Vitamin D Photoisomers From UVB-exposed Button Mushrooms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Gabriele Stangl, Prof. Dr., Martin-Luther-Universität Halle-Wittenberg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UHalle 2022-123
Record Dates: First submitted 2022-12-15; First posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Dietary Exposure; Safety Issues
Keywords: lumisterol; tachysterol; hydroxy-photoisomers; vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oral intake of UVB-exposed mushrooms (Experimental): Daily intake of 500 g of UVB-exposed button mushrooms over 7 days (provided as mushroom cream soup) and blood sampling (at baseline, 3 h postprandial, 6 h postprandial and at day 8)
  Interventions: Dietary Supplement: UVB-exposed button mushrooms
- oral intake of non-UVB-exposed mushrooms (Placebo Comparator): Daily intake of 500 g of non-UVB-exposed button mushrooms over 7 days (provided as mushroom cream soup) and blood sampling (at baseline, 3 h postprandial, 6 h postprandial and at day 8)
  Interventions: Dietary Supplement: UVB-exposed button mushrooms

INTERVENTIONS:
Dietary Supplement: UVB-exposed button mushrooms — Healthy subjects will be randomized into two groups and received either UVB-exposed button mushrooms or non-UVB-exposed button mushrooms for 7 days. Blood samples from each subject will be taken at baseline (before the intake of the mushrooms, 3 h and 6 h thereafter, and at day 8. Three months later, another blood sample was taken.

SUMMARY:
The European Food Safety Authority has approved many applications for UVB light treated foods (e.g. UVB-exposed button mushrooms) in the last years. The UVB light treatment is used to increase the vitamin D content in foods and improve the vitamin D status of subjects. However, UVB irradiation is accompanied by the formation of vitamin D photoisomers such as lumisterol and tachysterol. The current study aims to investigated whether these vitamin D photoisomers can enter the circulation and are metabolised in humans that consume UVB-treated mushrooms.

DETAILED DESCRIPTION:
according to protocol

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Age between 18 and 65 years
* Body Mass Index in the range of 18.5 to 29.9 kg/m2

Exclusion Criteria:

* Acute or chronic illnesses (high blood pressure, heart disease, diabetes, kidney disease, liver disease, alcohol dependence, etc.)
* Taking medication (except oral contraceptives)
* Pregnancy or breastfeeding
* Food intolerances or allergies to mushrooms and dairy products
* Smokers
* Visits to solariums or previous holidays in southern countries or in the Alps or other high mountains
* Participation in another study
* Blood donation during the last 2 months before the start of the study
* Dieting
* Severe weight loss or weight loss (≥ 3 kg) within the last month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-01-09 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Circulating vitamin D photoisomers | at baseline (before the intervention), 3 hours postprandial, 6 hours postprandial, at day 8, changes from baseline at 3 months
  Plasma concentrations of vitamin D photoisomers (such as lumisterol, tachysterol and their hydroxy derivates) after the consumption of the UVB-exposed versus non UVB-exposed button mushrooms

SECONDARY OUTCOMES:
Parameters of vitamin D metabolism | at baseline (before the intervention), 3 hours postprandial, 6 hours postprandial, at day 8, changes from baseline at 3 months
  Plasma concentrations of vitamin D metabolites (vitamin D2, vitamin D3, 25-hydroxyvitamin D2, 25-hydroxyvitamin D3, 24,25-dihydroxyvitamin D2, calcitriol, ergosterol)
Parameters of mineral metabolism | at baseline (before the intervention), 3 hours postprandial, 6 hours postprandial, at day 8, changes from baseline at 3 months
  Plasma calcium, phosphate, parathyroid hormone, fibroblast growth factor-23
Plasma lipids | at baseline (before the intervention), 3 hours postprandial, 6 hours postprandial, at day 8, changes from baseline at 3 months
  Plasma triglycerides, cholesterol
Inflammation markers | at baseline (before the intervention), 3 hours postprandial, 6 hours postprandial, at day 8, changes from baseline at 3 months
  Plasma CRP, Interleukin-6
mRNA and protein expression in peripheral mononuclear blood cells | at baseline (before the intervention), 3 hours postprandial, 6 hours postprandial, at day 8, changes from baseline at 3 months
  Vitamin D receptor target genes, CYP enzymes

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele I Stangl, Prof. Dr., Principal Investigator — Martin-Luther-Universität Halle-Wittenberg